CLINICAL TRIAL: NCT01768455
Title: A Randomized, Open Label Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Gemigliptin and Glimepiride in Healthy Male Subjects
Brief Title: Pharmacokinetic Drug Interaction Study Between Gemigliptin and Glimepiride in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL013
Record Dates: First submitted 2013-01-13; First posted 2013-01-15 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444; glimepiride

ARMS (2):
- Gemigliptin and Glimepiride (Experimental): Multiple administrations of gemigliptin and single concomitant administration of gemigliptin and glimepiride
  Interventions: Drug: Gemigliptin and Glimepiride
- Glimepiride (Experimental): Single administration of glimepiride
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Gemigliptin and Glimepiride — Gemigliptin 50mg (qd) on Day1~Day6 and Gemigliptin 50mg (qd) and Glimepiride 4mg (qd) on Day7
  Arms: Gemigliptin and Glimepiride
Drug: Glimepiride — Glimepiride 4mg (qd) on Day1
  Arms: Glimepiride

SUMMARY:
The objective of the study was to investigate the pharmacokinetic drug interaction between gemigliptin and glimepiride in healthy male subjects after oral administration concomitantly and each alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45, healthy male subjects (at screening)
* BMI between 18 - 27 (at screening)
* FPG 70-125mg/dL glucose level (at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(gemigliptin, glimepiride, aspirin, antibiotics)
* Subject who already participated in other trials in 90 days
* Subject who had whole blood donation in 60 days, or component blood donation in 30 days or transfusion in 30 days currently

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
AUC | up to 24h post-dose
  To evaluate AUCτ,ss of gemigliptin and AUClast of glimepiride
Cmax | up to 24h post-dose
  To evaluate Cmax,ss of gemigliptin and Cmax of glimepiride

SECONDARY OUTCOMES:
Tmax | up to 24h post-dose
  To evaluate Tmax,ss of gemigliptin/LC15-0636 and Tmax of glimepiride/M1
t1/2β | up to 24h post-dose
  To evaluate t1/2β of gemigliptin/LC15-0636/glimepiride/M1
AUC | up to 24h post-dose
  To evaluate AUCτ,ss of LC15-0636 and AUClast of M1
Cmax | up to 24h post-dose
  To evaluate Cmax,ss of LC15-0636 and Cmax of M1

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea